CLINICAL TRIAL: NCT00675909
Title: Improving Sedation of Children Undergoing Procedures in the Emergency Department: Evaluation of Different Dosages and Routes of Administration of the Sedative Midazolam
Brief Title: Improving Sedation of Children Undergoing Procedures in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Eileen Klein, Professor, Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2005-0260A
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Results first posted 2012-06-07 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Anxiety
Keywords: Sedation; Anxiety; Minor procedures; Emergency Department
MeSH Terms: conditions — Anxiety Disorders; Emergencies | interventions — Midazolam

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oral Midazolam (Active Comparator): Oral midazolam 0.5mg/kg
  Interventions: Drug: Oral midazolam
- Aerosolized intranasal midazolam (Experimental): Intranasal midazolam 0.3mg/kg
  Interventions: Drug: Aerosolized Intranasal midazolam
- Aerosolized buccal midazolam (Experimental): Buccal midazolam 0.3mg/kg
  Interventions: Drug: Aerosolized Buccal Midazolam

INTERVENTIONS:
Drug: Aerosolized Intranasal midazolam — Midazolam will be administered via aerosolization (using "atomizer") with half of dose in each nostril. Total dose is 0.3mg/kg.
  Other Names: Versed
  Arms: Aerosolized intranasal midazolam
Drug: Aerosolized Buccal Midazolam — 0.3mg/kg total dose administered with aerosolization device ("atomizer") sprayed onto buccal mucosa inside the cheek on both sides of mouth.
  Other Names: Versed
  Arms: Aerosolized buccal midazolam
Drug: Oral midazolam — oral midazolam 0.5mg/kg
  Other Names: Versed
  Arms: Oral Midazolam

SUMMARY:
Lacerations (deep cuts) are a frequent cause of visits to emergency departments and laceration repair is one of the most common procedures performed in that setting. Children are often anxious when they visit the emergency department, and visits where they anticipate needing painful procedures can be particularly stressful. Though we can manage the pain associated with many minor procedures, we are frequently unable to adequately support the child and treat their problem if we don't manage their anxiety as well. Methods of calming that do not require medication (e.g. distraction, parental support) can help, but many patients still require sedative medications.

The goal of sedation in the pediatric emergency department is to relieve the child's anxiety while minimizing the risk of adverse events. Unfortunately, when sedative medications are used in doses that do not slow breathing, they often fail to manage the child's anxiety adequately. In addition, many sedative agents require the placement of an intravenous line, which is itself a painful procedure that can create, rather than relieve, anxiety.

Currently, there is no ideal sedative agent that is safe, effective, and easy to administer. Oral midazolam is one of the most commonly used sedative medications for laceration repair in children. In a dose of 0.5mg/kg it has been shown to be safe. Unfortunately, it provides adequate sedation in only about two thirds of patients and has a delayed onset of up to 20 minutes. The remaining children must either endure the procedure in an agitated state or suffer placement of an intravenous line to administer additional sedative medications.

We aim to find a method of providing sedation for laceration repair that has a higher success rate than oral midazolam as currently prescribed without increasing the risk of complications. We would like to evaluate new methods for administering midazolam using alternate routes and dosages. Previous studies have looked at the use of midazolam absorbed directly by mucous membranes such as inside the nose (intranasal) and inside the mouth (buccal). The use of intranasal midazolam has had some success especially given its rapid onset of action (about 5 minutes), but has been limited by the irritant effects of the drug. When placed in the mouth, many children swallow the drug or spit it out rather than allowing it to be absorbed by the mucous membrane. There has been some improved success when the drug was placed under the tongue, but this is typically difficult for young children. However, a new device called an "atomizer" has been developed that allows for improved intranasal and buccal administration. The "atomizer" has a small adapter placed on the end of a syringe, which spreads the medication out in a fine mist over a wide area. It can be sprayed in the mouth inside the cheek (buccal), avoiding the need to keep the medication under the tongue. While some pediatric institutions have already started giving midazolam with the atomizer, and are reporting anecdotal success with these methods, its safety and effectiveness have not been rigorously studied.

We propose to compare three approaches to sedation: commonly used doses of oral midazolam, atomized intranasal midazolam and atomized intraoral midazolam. Children under the age of 7 requiring sedation for wound repair will be eligible for enrollment. After informed consent, children will be randomized to one of the three methods described above. Their level of sedation will be determined using two scores validated for use in children (the sedation score and the modified CHEOPS score). Physician, nurse and parent impressions of sedation will also be compared.

By comparing our current approach to these new methods, we will be able to determine which method is best. If we can identify a method for administering the sedative drug midazolam that is safe, well tolerated, and more effective, we will have made a valuable and important contribution to the care of injured children in the emergency department.

DETAILED DESCRIPTION:
The goal of this study is to improve sedation of children undergoing laceration repair in the emergency department. Currently, children who require sedation for laceration repair most often receive short acting benzodiazepines (i.e.,midazolam) orally (by mouth). Studies on the effectiveness of oral midazolam for minor procedures cite a 50-75% success rate. Oral midazolam has variable effectiveness and onset of action, and due to first pass hepatic metabolism, oral midazolam has a bioavailability of only 27% in children (Blumer 1998). Given the low success rate of oral midazolam, administration via mucous membranes has also been attempted. When administered intranasally or buccally, midazolam has a much higher bioavailability (Walberg 1991) and more rapid onset of action. Unfortunately, when given by these routes in previous studies, it was dripped into the nose or placed under the tongue. This leads to either swallowing the liquid drug, or expelling it, leading again to suboptimal bioavailability. Moreover, intranasal midazolam is irritating to the nasal mucosa and has therefore not always been well tolerated. When given to cooperative adults, midazolam dripped onto mucosal surfaces can have a bioavailability of approximately 75% (Schwagmeier 1998).

It has been hypothesized that better distribution of midazolam on mucosal surfaces would improve the reliability and effectiveness of this route of administration. A device called an atomizer has been developed for just this purpose (Wolfe Tory Medical, Inc., Salt Lake City, UT). The atomizer is an attachment on the end of a small syringe that causes the medication to be propelled over a larger surface area in a spray (see Figure below). This allows a greater percentage of the medication to be absorbed via the mucosal surface with a direct route to the blood stream leading to faster and more reliable onset of action, while avoiding the problem of hepatic metabolism that occurs with enterally absorbed midazolam.

We propose a study to determine if changes in the mode of administration and dosing of midazolam can provide improved sedation for children undergoing anxiety-producing procedures, without adversely effecting safety, length of stay, or patient/family and staff satisfaction.

To study this, we propose a randomized clinical trial to compare three methods of administering midazolam for sedation: oral midazolam 0.5 mg per kg, buccal midazolam 0.3 mg per kg and intranasal midazolam 0.3 mg per kg. The subject population will be children under the age of 7 who require sedation for laceration repair in the Emergency Department of Children's Hospital and Regional Medical Center. Patients will be excluded if they have: closed head injury with loss of consciousness, abnormal neurologic exam relative to baseline status, severe developmental delay or baseline neurologic deficits, severe trauma with suspected internal injuries, acute or chronic respiratory conditions, or renal, cardiac or hepatic abnormalities.

Variables of interest will include level of sedation prior to and during the procedure (using an activity scale and a modified CHEOPS scale) (McGrath 1985), time to adequate sedation, procedure length, length of ED stay, parental, MD, and RN satisfaction using a Likert scale, and complications such as respiratory depression and vomiting as well as measures needs to ameliorate those complications. For adequate power, we anticipate enrolling 180 patients (60 in each treatment group) during the 24-month duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Laceration in need of repair with sutures, with no other major injuries
2. Age >=6 months and < 7 years
3. No meal within the last 2 hours

Exclusion Criteria:

1. Closed head injury associated with loss of consciousness
2. Abnormal neurologic exam, relative to baseline status
3. Significant developmental delay or baseline neurologic deficit
4. Severe trauma with suspected internal injuries
5. Acute or chronic respiratory condition
6. Acute or chronic renal, cardiac or hepatic abnormalities
7. Allergy to benzodiazepines or previous reaction to benzodiazepines
8. Taking erythromycin containing antibiotics
9. Nasal and intraoral lacerations

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2006-11; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen J Klein, MD, MPH, Principal Investigator — Associate Professor, Pediatrics

REFERENCES:
- [Result] Klein EJ, Brown JC, Kobayashi A, Osincup D, Seidel K. A randomized clinical trial comparing oral, aerosolized intranasal, and aerosolized buccal midazolam. Ann Emerg Med. 2011 Oct;58(4):323-9. doi: 10.1016/j.annemergmed.2011.05.016. PMID 21689865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment November 2006-January 2010 from the Emergency Department at Seattle Children's Hospital
Groups:
- Oral Midazolam: Participants in the group are given oral midazolam as sedation related to laceration repair procedures in the emergency department.
  0.5mg/kg of midazolam taken orally.
- Buccal Midazolam: Participants in the group are given buccal midazolam as sedation related to laceration repair procedures in the emergency department.
  0.3mg/kg total dose administered with aerosolization device ("atomizer") sprayed onto buccal mucosa inside the cheek on both sides of mouth.
- Intranasal Midazolam: Participants in the group are given intranasal midazolam as sedation related to laceration repair procedures in the emergency department.
  Midazolam will be administered via aerosolization (using "atomizer") with half of dose in each nostril. Total dose is 0.3mg/kg.
Period: Overall Study
Arm/Group | Oral Midazolam | Buccal Midazolam | Intranasal Midazolam
Started | 60 | 60 | 60
Completed | 60 | 60 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Midazolam | Buccal Midazolam | Intranasal Midazolam | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 60 | 60 | 180
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.1 (1.5) | 3.7 (1.4) | 3.2 (1.3) | 3.3 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 20 | 20 | 67
  Male | 33 | 40 | 40 | 113
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 60 | 180

OUTCOME MEASURES:

1. Primary Outcome: Change in CHEOPS Score Measured Level of Sedation From Baseline (Presentation in ED, Before Sedation) to Start of Procedure (Laceration Repair).
Description: Modified CHEOPS (Children's Hospital of Eastern Ontario Pain Scale)assessment used to score sedation.
  Scale range is 0-10 with 0 meaning no pain and 4 or greater meaning pain. Scale is determined by assessing Facial Expression (0-2), Cry (0-3), Child Verbal (0-2) and Movements (0-3).
Time Frame: Baseline (presentation, before sedation) in ED to start of procedure (laceration repair).
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Oral Midazolam | Intranasal Midazolam | Buccal Midazolam
Number analyzed (Participants) | 56 | 55 | 58
Scores on a scale | 2 [-2 to 7] | 2 [-3 to 7] | 1 [-6 to 6]

2. Secondary Outcome: Time From Study Drug Administration to Start of Procedure
Time Frame: Time from study drug administration to start of procedure up to 68 minutes
Measure: Median (Full Range); unit: minutes
Arm/Group | Oral Midazolam | Intranasal Midazolam | Buccal Midazolam
Number analyzed (Participants) | 58 | 55 | 58
minutes | 34 [11 to 68] | 28 [5 to 60] | 32 [10 to 59]

3. Secondary Outcome: Duration of Procedure
Time Frame: Duration of procedure up to 40 minutes
Measure: Median (Full Range); unit: minutes
Arm/Group | Oral Midazolam | Intranasal Midazolam | Buccal Midazolam
Number analyzed (Participants) | 58 | 54 | 58
minutes | 12 [1 to 40] | 12 [1 to 40] | 10 [1 to 39]

4. Secondary Outcome: Physician Rating of Sedation
Description: Range is 0-10. Higher is associated with physician impression that sedation is better.
Time Frame: Physician was asked after the procedure was done about their impression of sedation.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Oral Midazolam | Intranasal Midazolam | Buccal Midazolam
Number analyzed (Participants) | 57 | 52 | 58
units on a scale | 6.7 [0 to 10] | 8.1 [1 to 10] | 7.1 [0 to 10]

5. Secondary Outcome: Nurse Rating of Sedation
Description: Range is 0-10. Higher is associated with nurse impression that sedation is better.
Time Frame: After the procedure nurse was asked about their impression of the level of sedation.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Oral Midazolam | Intranasal Midazolam | Buccal Midazolam
Number analyzed (Participants) | 43 | 44 | 44
units on a scale | 6.8 [0 to 10] | 7.7 [1 to 10] | 7.6 [0 to 10]

ADVERSE EVENTS:
Arm/Group | Oral Midazolam | Buccal Midazolam | Intranasal Midazolam
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes